CLINICAL TRIAL: NCT00358241
Title: Effects of Continuous Lumbar Plexus Nerve Block on Functional Restoration and Outcome After Unilateral Total Knee Arthroplasty
Brief Title: Effects of Nerve Block on Knee Function After Knee Replacement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left JHU and is not able to be reached for updates
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 04-03-05-05
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2019-05

CONDITIONS: Postoperative Pain
Keywords: Nerve block, postoperative pain, analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Nerve Block

INTERVENTIONS:
Procedure: Nerve block

SUMMARY:
Early physical therapy after knee surgery is very painful on top of pain from surgery. Pain following surgery can limit recovery. One way to treat pain is by giving intravenous (IV) pain medication with morphine. Another method is to use a "nerve block" which involves placing a thin catheter (tube) into the lower back near the nerves that sense pain in the knee and give a local anesthetic to numb the nerves. Sometimes both methods are used together. This research is being done to determine whether nerve blocks with a local anesthetic improve knee recovery in addition to providing pain relief as compared to IV pain medicine alone

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80 year old
* ASA Physical Status ASA I and II
* Mentally competent
* Intellectually competent
* Body mass index <35
* No severe cardiac diseases
* No severe pulmonary diseases
* Unilateral knee disease
* No other lower extremity joint disease
* No chronic narcotic therapy or illicit drug use

Exclusion Criteria:

* Age <21 or >80 year old
* ASA Physical Status >ASA II
* Mentally incompetent
* Intellectually incompetent or cognitively impaired
* Non-English speaking patient
* Worker's compensation patient
* Body mass index > 35
* Bilateral knee disease
* Has other lower extremity joint disease
* Severe cardiac diseases
* Severe pulmonary diseases
* Chronic narcotic therapy or illicit drug use
* Pregnancy

Ages: 21 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Hang, MD, PhD, Principal Investigator — Johns Hopkins Medicine, Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States